CLINICAL TRIAL: NCT02226068
Title: Ciclosporine and Extracorporal Photopheresis (ECP) Are Equipotent in Treating Severe Atopic Dermatitis (AD): A Randomized Cross-over Study Comparing Two Efficient Treatment Modalities
Brief Title: Photophoresis Versus Ciclosporine in Severe Atopic Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Purpose: Treatment
Other Study IDs: CsAvsECP-AUH; CsA-ECP (Other: DermatologyAUH-UK)
Record Dates: First submitted 2014-08-25; First posted 2014-08-26 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2014-08

CONDITIONS: Atopic Dermatitis
Keywords: Atopic dermatitis; Ciclosporine; Extracorporal photopheresis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Cyclosporine; Photopheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CsA-ECP (Other): Sequence of therapy: First ciclosporin was given and after relapse extra corporal photopheresis was given
  Interventions: Drug: Cyclosporine A (CsA); Other: Extracorporeal photopheresis (ECP)
- ECP-CsA (Other): Sequence of therapy: First extra corporal photopheresis was given and after relapse ciclosporin was given
  Interventions: Drug: Cyclosporine A (CsA); Other: Extracorporeal photopheresis (ECP)

INTERVENTIONS:
Drug: Cyclosporine A (CsA) — 3 mg/kg/day for 4 month
  Other Names: Sandimmune
Other: Extracorporeal photopheresis (ECP) — Administered two consecutive days twice a month for 4 month

SUMMARY:
Severe atopic dermatitis (AD) is a recurrent and debilitating disease often requiring systemic immunosuppressive treatment. The efficacy of cyclosporine A (CsA) is well proven but potential side effects are concerning. Several reports point at extracorporeal photopheresis (ECP) as an efficient alternative treatment modality with few and mild side effects. However, no direct comparison between CsA and ECP in the treatment of AD has been performed so far. In this trial we test the hypothesis that ECP is non-inferior to standard treatment with CsA.

ELIGIBILITY:
Inclusion Criteria:

Criteria of inclusion were refractoriness to standard topical treatment (corticosteroid ointments, UVA, UVB, PUVA, tar).

Exclusion Criteria:

Criteria of exclusion were pregnancy, uncontrolled hypertension, previous malignancy, infectious disease, liver/kidney disease or active treatment with ECP or immunosuppressants within 4 weeks prior to start of trial.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2002-06; Primary Completion 2003-08 (Actual); Study Completion 2004-01 (Actual)

PRIMARY OUTCOMES:
Change of SCORAD (SCORing Atopic Dermatitis) | 4 month

CONTACTS AND LOCATIONS:
Overall Officials: Erik Obitz, MD, DMSc, Principal Investigator — Department of Dermatology, Aarhus University Hospital, Aarhus, Denmark